CLINICAL TRIAL: NCT03876236
Title: Danish Anaesthesia Study (DANA) 0: Reproducibility of Structural and Functional Magnetic Resonance Imaging of the Brain in Healthy Volunteers - a Pilot Study. First Substudy of the Protocol, 'Neuroplasticity Induced by General Anaesthesia'
Brief Title: Reproducibility of Brain MRI
Acronym: DANA0
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kirsten Moller, Professor, MD, consultant, PhD, DMSc, Rigshospitalet, Denmark
Other Study IDs: H-18020364
Record Dates: First submitted 2019-02-08; First posted 2019-03-15 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Reproducibility of Results
Keywords: Magnetic Resonance Imaging; Diffusion Tensor Imaging; Reproducibility of Results; Feasibility Study; Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rest: Quiet rest in supine position, 2 hrs.

SUMMARY:
The aim of this study is to assess the reproducibility over time of functional and structural magnetic resonance imaging, as well as specific biomarkers in plasma in healthy volunteers before and after a two-hour rest. This design mimics the timing of repeated scans and blood sampling before and after two hours of anaesthesia in subsequent substudies of the protocol, 'Neuroplasticity Induced by General Anaesthesia'.

DETAILED DESCRIPTION:
In the study 'Neuroplasticity Induced by General Anaesthesia', the investigators intend to explore the effects of general anaesthesia on the brain by state-of-the-art magnetic resonance imaging (MRI).

MRI data - especially changes in functional MRI recordings - may theoretically depend on a variety of physiological variables such as cerebral blood flow, cerebral blood volume, and cerebral metabolic oxidative rate of oxygen, and may thus also be affected by pharmacological agents. However, to interpret data it is important to know the inherent variability of the scans.

This first substudy therefore aims to determine the reproducibility of the MRI recordings without administration of pharmacological agents. Another aim of the study is to ensure feasibility of the design before embarking on the more resource-demanding substudies in anaesthetised subjects.

In this substudy, the investigators will perform the same MRI measurements as in the main study; rather than undergoing two hours of general anaesthesia, the volunteers will be subjected to two hours of undisturbed rest.

Each participant goes through a pre-study interview and physical examination to ensure that the participant is healthy and suitable for participation.

For each participant, the study consists of three study days:

Day 0: Baseline MRI and blood tests. Intervention. Two hours of post-intervention care followed by post-intervention MRI and blood tests.

Day +1 (the day after Day 0): MRI and blood tests. Day +7 (one week after Day 0): MRI and blood tests.

All MRI scans will be performed with a 3 Tesla Philips Achieva d-stream with a 32-channel receive head coil.

Blood tests: Haemoglobin, sodium, potassium, white blood count, C-reactive protein (CRP), S calcium-binding protein 100b (S100b), neuron-specific enolase (NSE), interleukin-1 (IL-1), IL-6, IL-8, IL-10, IL-18, tumor necrosis factor Alpha (TNF-Alpha) and transforming growth factor beta (TGF-beta).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 ≤35
* Healthy individual
* Normal electrocardiogram (ECG)
* Normal physical examination, including neurological examination, auscultation of the heart and lungs, and measurement of blood pressure and pulse.
* Speaks and understands Danish
* Provides oral and written informed consent
* Right-handed
* American Society of Anaesthesiologists (ASA) class 1 (2)
* Mallampati I-II and simplified airway risk index (SARI) 0-2 (i.e. no indication of difficult intubation. See Appendix for details)
* BMI ≥18 kg/m2 and ≤30kg/m2
* Female participants must use safe contraceptives.

Exclusion Criteria:

* Cannot cooperate to tests
* Left-handedness or ambidexterity
* History of cancer, immune disease, autoimmune disease, chronic pain, neurological / psychiatric illness or other serious illness
* Pregnancy
* Weakly intake of >21 (males) or >14 (females) units of alcohol
* Substance abuse (assessed by the investigator)
* Daily use of any medication (contraceptives allowed)
* Consumed anti-depressants during the last 30 days before study days
* Heavy intake of caffeine (> 5 cups/day)
* Smoking during the last 30 days before study days
* Reflux or dyspepsia
* Poor dental status or oral health
* Contraindication to MRI
* Allergy to any kind of medication or material to which the volunteer could be exposed to during this study
* Family history of malignant hyperthermia
* Declines receiving information regarding incidental pathological findings during MRI scans of the brain.
* Otherwise judged unfit for participation by the investigator
* Major trauma or head trauma with any symptoms present at the time of inclusion
* Surgery less than six weeks prior to the study period
* Infection (with fever) less than two weeks prior to the study period
* Expected or suspected difficult airway
* History of complications to general anaesthesia
* Known incident of malignant hyperthermia or unexplained complications to general anaesthesia among close relatives.

Exclusion criteria during the study (leading to withdrawal):

* Any of the above-mentioned exclusion criteria
* Consumption of more than 3 units of alcohol within 24 hours before each study day (intervention day or MRI scan day)
* Consumed analgesics within 3 days before each study day
* Consumed anti-histamines less than 48 hours before each study day
* Intake of caffeine 12 h prior to each study day
* Smoking
* Major trauma or head trauma during the study period
* Surgery less during the study period
* Fever due to any infection < 14 days before the study or during the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young volunteers
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Feasibility and reproducibility: rates of protocol violation and delays as well as adverse events | 8 days
  Evaluation of feasibility of study set-up, as measured by rates of protocol violation and delays as well as adverse events. The time frame mentioned below runs from the first study day, NOT from eligibility interview.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Moller, MD PhD MDSc, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Neuroanaesthesiology, Glostrup Municipality, Capital Region
  - Functional Imaging Unit, Department for Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet Glostrup, Glostrup Municipality, Capital Region

IPD SHARING:
Plan to Share IPD: No
The responsible investigators will consider data sharing, considered compliance with GDPR regulations and data sharing agreement.